CLINICAL TRIAL: NCT03532074
Title: Intraoperative Assessment of Bowel Perfusion Through Indocyanine Green in Women With Rectosigmoid Endometriosis and Its Correlation With Clinical and Surgical Data
Brief Title: Indocyanine Green and Rectosigmoid Endometriosis
Acronym: vincendo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Mohamed Mabrouk, Principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 290/2017/O/Sper
Record Dates: First submitted 2018-04-09; First posted 2018-05-22 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Endometriosis, Rectum; Bowel Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Masking Description: OPEN
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic approach (Other): assessment of bowel symptoms before surgery; assessment of rectosigmoid perfusion using indocyanine green; removal of rectosigmoid endometriosis nodule using a laparoscopic approach; follow up and assessment of bowel symptoms after surgery
  Interventions: Diagnostic Test: assessment of bowel symptoms before surgery; Diagnostic Test: assessment of rectosigmoid during laparoscopy; Diagnostic Test: follow up and assessment of bowel symptoms after surgery
- robot-assisted approach (Other): assessment of bowel symptoms before surgery; assessment of rectosigmoid perfusion using indocyanine green; removal of rectosigmoid endometriosis nodule using a robot-assisted approach; follow up and assessment of bowel symptoms after surgery
  Interventions: Diagnostic Test: assessment of bowel symptoms before surgery; Diagnostic Test: follow up and assessment of bowel symptoms after surgery; Diagnostic Test: assessment of rectosigmoid perfusion during robot-assisted laparoscopy

INTERVENTIONS:
Diagnostic Test: assessment of bowel symptoms before surgery — validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire and Gastrointestinal Quality of Life Index) are filled in by patients with rectosigmoid endometriosis before surgery
Diagnostic Test: assessment of rectosigmoid during laparoscopy — indocyanine green (0.25 mg/kg) is administered through peripheral line. A near-infrared camera-head (KARL STORZ Gesellschaft mit beschränkter Haftung & Co., Tuttlingen, Germany) is used to visualize bowel perfusion before and after the removal of the rectosigmoid nodule. To estimate the vascularization, a scale with a score between 0 and 4 is used
  Arms: laparoscopic approach
Diagnostic Test: follow up and assessment of bowel symptoms after surgery — validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire and Gastrointestinal Quality of Life Index) are filled in by patients with rectosigmoid endometriosis after surgery
Diagnostic Test: assessment of rectosigmoid perfusion during robot-assisted laparoscopy — indocyanine green (0.25 mg/kg) is administered through peripheral line. The robotic Firefly imaging system (daVinciXi surgical platform; Intuitive Surgical, Sunnyvale, CA) is used to visualize bowel perfusion before and after the removal of the rectosigmoid nodule. To estimate the vascularization, a scale with a score between 0 and 4 is used
  Arms: robot-assisted approach

SUMMARY:
Indocyanine green is a fluorescent dye used for the intraoperative evaluation of tissue perfusion.

The aim of this study is to evaluate a possible correlation between rectosigmoid vascularization and surgical and clinical data including pre and post-operative bowel symptoms in patients needing surgery for rectosigmoid endometriosis.

DETAILED DESCRIPTION:
Patients with symptomatic rectosigmoid endometriosis requiring laparoscopic surgery are included in the study.

Before surgery, bowel symptoms are assessed using validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire and Gastrointestinal Quality of Life Index).

Indocyanine green is administered through peripheral line. A near-infrared (NIR) camera-head enables real-time direct visualization of bowel perfusion before and after the removal of the rectosigmoid nodule. Rectosigmoid tract perfusion is assessed before and after the removal of the nodule. To estimate the vascularization, a scale with a score between 0 and 4 is used.

After complete removal of rectosigmoid nodule, the post-operative follow-up will be the same as usual after intestinal endometriosis surgery. Postoperative bowel symptoms are evaluated using the same questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of deep endometriosis based on clinical and transvaginal/transabdominal ultrasound examinations and, when necessary, magnetic resonance
* Patients with indication for removal of endometriosic lesions by laparoscopic surgery
* Obtaining Informed Consent

Exclusion Criteria:

* Known or suspected allergy to iodine
* Previous rectal surgery
* History of active pelvic infection
* Intra-abdominal or pelvic malignancy
* Pelvic radiation therapy
* Hyperthyroidism
* Liver dysfunction
* Serum creatinine > 2.0 mg/dL

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
correlation between bowel symptoms and rectosigmoid perfusion before the nodule removal | intraoperative
  comparison between bowel symptoms, assessed through validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire and Gastrointestinal Quality of Life Index) and rectosigmoid perfusion, measured before the nodule removal using indocyanine green and a scale from 0 to 4.

SECONDARY OUTCOMES:
correlation between bowel symptoms and rectosigmoid perfusion after the nodule removal | up to three months after surgery
  comparison between rectosigmoid perfusion, measured after the nodule removal using indocyanine green and a scale from 0 to 4, and bowel symptoms, assessed through validated questionnaires (Knowles-Eccersley-Scott-Symptom Questionnaire and Gastrointestinal Quality of Life Index).
correlation between bowel perfusion after rectal surgery and post-operative complications | up to three months after surgery; from date of surgery until the date of first documented complication, assessed up to 3 months
  assessment of rectosigmoid perfusion, through indocyanine green and a scale from 0 to 4, and complications (rectovaginal fistula, dehiscence of anastomotic suture, rectal bleeding, rectosigmoid perforation, rectosigmoid stenosis), using Clavien-Dindo Classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology and Physiopathology of Human Reproductive Unit, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy